CLINICAL TRIAL: NCT02481947
Title: A Safety and Efficacy Evaluation of BLI400 Laxative in Constipated Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLI400-301
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BLI400 Laxative (Experimental): 21 gm BLI400 powder
  Interventions: Drug: BLI400 Laxative
- Lubiprostone (Active Comparator): 24 mcg capsule bid
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: BLI400 Laxative — 21 gm BLI400 powder
  Arms: BLI400 Laxative
Drug: Lubiprostone — 24 mcg capsule bid
  Arms: Lubiprostone

SUMMARY:
The purpose of this study is to evaluate a daily dose of BLI400 Laxative for safety and efficacy versus lubiprostone in constipated adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age
* Constipated, defined by the following adapted ROME II definition:

A. Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for at least 12 weeks (which need not be consecutive) in the preceding 12 months:

1. Straining during > 25% of defecations
2. Lumpy or hard stools in > 25% of defecations
3. Sensation of incomplete evacuation for > 25% of defecations

B. Loose stools are rarely present without the use of laxatives

C. There are insufficient criteria for IBS - loose (mushy) or watery stool in the absence of laxative use for more than 25% of bowel movements

Criteria A, B and C must be fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.

* Otherwise in good health, as determined by physical exam and medical history
* If female, and of child-bearing potential, is using an acceptable form of birth control
* Negative urine pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
* Subjects who have had major surgery 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
* Subjects with hypothyroidism that is being treated and for which the dose of thyroid hormone has not been stable for at least 6 weeks at the time of Visit 1
* Subjects taking laxatives, enemas or prokinetic agents that refuse to discontinue these treatments from Visit 1 until after completion of Visit 5
* Subjects who are pregnant or lactating, or intend to become pregnant during the study
* Subjects of childbearing potential who refuse a pregnancy test
* Subjects who are allergic to any study medication component
* Subjects taking narcotic analgesics or other medications known to cause constipation
* Subjects with clinically significant cardiac abnormalities identified at the Visit 1 ECG
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
* Subjects with an active history of drug or alcohol abuse
* Subjects have been hospitalized for a psychiatric condition or have made a suicide attempt during the 2 years before Visit 1
* Subjects who withdraw consent at any time prior to completion of Visit 1 procedures
* Subjects with known or suspected moderate to severe hepatic insufficiency (Child Pugh Classes B and C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (50):
- United States (50):
  - BLI Research Site 38, Mobile, Alabama
  - BLI Research Site 21, Tucson, Arizona
  - BLI Research Site 10, Anaheim, California
  - BLI Research Site 12, Artesia, California
  - BLI Research Site 28, Corona, California
  - BLI Research Site 30, La Mirada, California
  - BLI Research Site 13, Laguna Hills, California
  - BLI Research Site 41, Orange, California
  - BLI Research Site 50, Sacramento, California
  - BLI Research Site 23, San Diego, California
  - BLI Research Site 26, Brandon, Florida
  - BLI Research Site 4, Brandon, Florida
  - BLI Research Site 44, Clearwater, Florida
  - BLI Research Site 46, DeLand, Florida
  - BLI Research Site 32, Hialeah, Florida
  - BLI Research Site 40, Hialeah, Florida
  - BLI Research Site 5, Miami, Florida
  - BLI Research Site 34, Miami, Florida
  - BLI Research Site 36, Miami, Florida
  - BLI Research Site 8, Miami, Florida
  - BLI Research Site 17, Miami Lakes, Florida
  - BLI Research Site 43, Miami Springs, Florida
  - BLI Research Site 11, Orlando, Florida
  - BLI Research Site 18, Orlando, Florida
  - BLI Research Site 37, Palmetto Bay, Florida
  - BLI Research Site 24, St. Petersburg, Florida
  - BLI Research Site 3, Tampa, Florida
  - BLI Research Site 1, West Palm Beach, Florida
  - BLI Research Site 7, Atlanta, Georgia
  - BLI Research Site 25, Snellville, Georgia
  - BLI Research Site 16, Chicago, Illinois
  - BLI Research Site 47, Owensboro, Kentucky
  - BLI Research Site 6, Monroe, Louisiana
  - BLI Research Site 31, West Monroe, Louisiana
  - BLI Research Site 49, Las Vegas, Nevada
  - BLI Research Site 27, New York, New York
  - BLI Research Site 39, Raleigh, North Carolina
  - BLI Research Site 14, Cincinnati, Ohio
  - BLI Research Site 22, Chattanooga, Tennessee
  - BLI Research Site 29, Knoxville, Tennessee
  - BLI Research Site 45, Memphis, Tennessee
  - BLI Research Site 19, Nashville, Tennessee
  - BLI Research Site 20, Austin, Texas
  - BLI Research Site 9, Austin, Texas
  - BLI Research Site 42, Carrollton, Texas
  - BLI Research Site 48, Channelview, Texas
  - BLI Research Site 2, Plano, Texas
  - BLI Research Site 35, Charlottesville, Virginia
  - BLI Research Site 15, Newport News, Virginia
  - BLI Research Site 33, Richland, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- BLI400 Laxative: BLI400 Laxative (21 gm BLI400 powder per day)
- Lubiprostone: Lubiprostone (24 mcg capsule bid)
Period: Overall Study
Arm/Group | BLI400 Laxative | Lubiprostone
Started | 230 | 229
Completed | 184 | 193
Not Completed | 46 | 36
Not completed — Withdrawal by Subject | 24 | 10
Not completed — Lost to Follow-up | 11 | 5
Not completed — Adverse Event | 6 | 11
Not completed — Physician Decision | 4 | 5
Not completed — Protocol Violation | 1 | 5

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- BLI400 Laxative: BLI400 Laxative
  BLI400 Laxative: Oral laxative
- Lubiprostone: Lubiprostone
  Lubiprostone: Oral laxative
- Total: Total of all reporting groups
Arm/Group | BLI400 Laxative | Lubiprostone | Total
Number analyzed (Participants) | 230 | 229 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.6) | 45.6 (14.6) | 45.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 179 | 366
  Male | 43 | 50 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 98 | 193
  Not Hispanic or Latino | 135 | 131 | 266
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 63 | 68 | 131
  White | 156 | 146 | 302
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 8 | 10
Region of Enrollment [Number; unit: participants]
  United States | 230 | 229 | 459

OUTCOME MEASURES:

1. Primary Outcome: Complete Spontaneous Bowel Movement (CSBM) Response
Description: The primary endpoint is based on the number of subjects who are weekly responders for at least 9 out of 12 weeks, with at least 3 of these weeks occurring in the last 4 weeks of treatment. A weekly responder is a subject who has ≥ 3 CSBMs and an increase from baseline of > 1 CSBM in that week.
Time Frame: 12 weeks
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Groups:
- BLI400 Laxative: BLI400 Laxative (21 gm BLI400 powder)
Arm/Group | BLI400 Laxative | Lubiprostone
Number analyzed (Participants) | 187 | 199
Participants | 47 | 56
Statistical Analysis 1: Comparison: BLI400 Laxative vs Lubiprostone; Test type: Non-Inferiority — Non-inferiority margin = 12.6% (pre-specified); p = 0.016, Chi-squared — The a priori threshold for statistical significance was 0.05

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Results for mortality, serious adverse events and other adverse events are based on the FDA agreed upon Safety Population (BLI400 n=225, lubiprostone n=229).
Arm/Group | BLI400 Laxative | Lubiprostone
All-Cause Mortality (participants affected / at risk) | 1/225 | 0/229
Serious Adverse Events (participants affected / at risk) | 2/225 | 1/229
Other Adverse Events (participants affected / at risk) | 26/225 | 15/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI400 Laxative (N=225) | Lubiprostone (N=229)
Cellulitis of legs (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
stomach ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI400 Laxative (N=225) | Lubiprostone (N=229)
diarrhea (Gastrointestinal disorders) | 11 | 12
flatulence (Gastrointestinal disorders) | 17 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.